CLINICAL TRIAL: NCT03372083
Title: A Single-arm Interventional Phase IV, Post-authorisation Study Evaluating the Safety of Pediatric Patients With Transfusional Hemosiderosis Treated With Deferasirox Crushed Film Coated Tablets
Brief Title: Safety Study of Crushed Deferasirox Film Coated Tablets in Pediatric Patients With Transfusional Hemosiderosis
Acronym: MIMAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670F2429; 2016-003482-25 (EudraCT Number)
Record Dates: First submitted 2017-11-21; First posted 2017-12-13 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Iron Overload
Keywords: Iron Chelation Therapy; Deferasirox; Asunra; Jadenu; Exjade; ICL 670; Pediatric
MeSH Terms: conditions — Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deferasirox (Experimental): Crushed deferasirox (ICL670) FCT for oral use daily. Deferasirox FCT dosing was based on subject's weight.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — Deferosirox was provided in tablet forms of 90, 180 and 360mg. Tablets were crushed in the home environment and administered by sprinkling the full dose on to soft food to be consumed immediately.
  Other Names: ICL670

SUMMARY:
This study employed a prospective, single-arm, global multi-center interventional open-label, non-randomized design to identify and assess safety profile of the crushed deferasirox FCT when administered up to 24 weeks in pediatric patients aged ≥2 to <6 years with transfusional hemosiderosis. The study was designed to enroll a minimum of 40 patients. Forty-four patients were treated and analyzed.

DETAILED DESCRIPTION:
The study included a screening period (from Day 0-14) with two visits at least 7 days apart to assess eligibility of patients that were chelation naïve or on a prior iron chelator treatment other than DFX. For Patients on DFX treatment prior to study entry only one screening visit (screening visit 1) were to occur to determine eligibility. Any current chelation therapy except deferasirox were to be discontinued to undergo a 5-day washout period prior to commencing a 24 week treatment period with crushed deferasirox FCT.

All patients were to have weekly visits for the first month to monitor renal function. Hepatic function were to be assessed biweekly during the first month. Thereafter, monthly safety assessments were to be performed, including the monitoring of serum ferritin values and trends in order to adapt patient treatment.

Eligibility, application of dosing standards and adjustments, as well as safety and serum ferritin assessments as specified in the protocol.

The planned duration of treatment was 24 weeks followed by a 30-day safety follow up.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients ≥2 to <6 years old diagnosed with transfusional hemosiderosis
2. Documented history of red blood cell transfusions
3. Written informed consent/assent before any study-specific procedures. The consent will be obtained from caregiver(s) or patient's legal representative. Investigators will also obtain assent of patients according to local, regional, or national regulations.
4. For patients on prior DFX: Serum ferritin (SF) >500 ng/mL, measured at screening visit 1 and requiring a DFX daily dose equivalent to FCT ≥ 7mg/kg/day.
5. For patients on a prior chelator other than DFX (e.g. deferiprone or deferoxamine) or chelation naive: Serum ferritin (SF) >1000 ng/mL measured at screening visits 1 and 2.

Key Exclusion Criteria:

1. Patients that receive more than one iron chelator at the same time as current iron chelation treatment. (Patients who have received combination therapy in their medical history but are currently being treated with a single ICT agent are eligible.)
2. Patients continuing on deferoxamine or deferiprone in addition to study treatment. (Patients switching to or continuing on deferasirox are eligible).
3. Unresolved adverse events if the patient was previously treated with deferiprone or deferoxamine or deferasirox.
4. Significant proteinuria as indicated by a urinary protein/creatinine ratio > 0.5 mg/mg in a non-first void sample urine measured at screening visit 1.
5. Serum creatinine > age adjusted ULN measured at any screening visit
6. Creatinine clearance below 90 mL/minute measured at any screening visit. Creatinine clearance using the Schwartz formula will be estimated from serum creatinine measured at each respective visit.
7. ALT and/or AST > 2.5 x ULN measured at screening visit 1.
8. Total bilirubin (TBIL) >1.5 x ULN measured at screening visit 1.
9. Patients with significant impaired GI function or GI disease that may significantly alter the absorption of oral deferasirox FCT (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
10. History of and/or laboratory evidence of active Hepatitis B or Hepatitis C (HBsAg in the absence of HBsAb OR HCV Ab positive with HCV RNA positive.
11. Liver disease with severity of Child-Pugh Class B or C.
12. History of hypersensitivity to any of the study drug or excipients.
13. Patients participating in another clinical trial or receiving an investigational drug.
14. Patients with a known history of HIV seropositivity.
15. Patients unwilling or unable to comply with the protocol.
16. History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
17. Significant medical condition interfering with the ability to partake in this study (e.g. uncontrolled hypertension, unstable cardiac disease not controlled by standard medical therapy, systemic disease: cardiovascular, renal, hepatic, etc.).
18. Female patients who reach menarche and they or their caregivers refuse pregnancy testing and/or if there is a positive pregnancy test result.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Novartis Investigative Site, Zagazig, Egypt
- Italy (3):
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Cagliari, ITA
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Hazmiyeh, Beyrouth, Lebanon
- Novartis Investigative Site, Muscat, Oman
- Thailand (2):
  - Novartis Investigative Site, Bangkok Noi, Bangkok
  - Novartis Investigative Site, Muang, Chiangmai
- Novartis Investigative Site, Dubai, United Arab Emirates
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 10 sites in 7 countries (one in Egypt, three in Italy, one in Lebanon, one in Oman, two in Thailand, one in the United Arab Emirates, and one in the United Kingdom).
Period: Overall Study
Arm/Group | Deferasirox
Started (All enrolled patients were included in both the full analysis set (FAS) and the safety set) | 44
Completed | 39
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.05 (1.056)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 27
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 36
  Asian | 8
Baseline Body Mass Index [Mean (Standard Deviation); unit: kilogram per square metre (kg/m^2)] | 16.40 (2.009)
Baseline iron chelation naive participants [Count of Participants; unit: Participants]
  Chelation naive = Yes | 10
  Chelation naive = No | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Selected Gastrointestinal Disorders up to 24 Weeks
Description: To assess the safety of crushed deferasirox FCT with respect to selected gastrointestinal (GI) disorders (esophagitis, stomatitis, mouth ulceration, gastric ulcers, haemorrhage, abdominal pain, diarrhea, nausea, and vomiting). Only descriptive analysis performed.
Time Frame: Baseline (Week 1 Day 1) up to Week 24, plus 30 day safety follow-up.
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
Participants
  Oesophagitis | 0
  Barrett's esophagitis | 0
  Stomatitis | 0
  Mouth ulceration | 0
  Gastric ulcer | 0
  Gastrointestinal haemorrhage | 0
  Abdominal pain | 2
  Diarrhoea | 4
  Nausea | 0
  Vomiting | 2

2. Secondary Outcome: Adverse Events Profile
Description: Analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event TEAEs and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters. Only descriptive analysis performed.
Time Frame: Baseline (Week 1 Day 1) up to Week 24, plus 30 day safety follow-up.
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
Participants
  On treatment-related AE | 22
  On treatment related SAE | 0
  On treatment Deaths | 0

3. Secondary Outcome: Number of Participants With Notable Changes in ECG Values From Baseline
Description: Safety measured by the notable post-baseline changes in ECG values (PR, QRS, QT, QTcF and HR intervals) compared to baseline. Baseline was defined as the last non-missing value on or prior to the first dose. Only descriptive analysis performed.
Time Frame: Baseline (Week 1 Day 1) up to Week 24, plus 30 day safety follow-up.
Population: Safety set. For each parameter, only patients with a value at both baseline and post baseline were to be included.
Measure: Number; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
Participants | 0

4. Secondary Outcome: Absolute Change From Baseline in Serum Ferritin (SF)
Description: Absolute change from baseline over time in SF values up to 24 weeks of treatment were to be provided. Only descriptive analysis performed.
Time Frame: Baseline (BL), Week 4, Week 8, Week 12, Week 16, EOT (Week 24)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
ug/L
  Baseline (BL) | 2152.7 (1039.06)
  Change from BL @ Week 4: number analyzed (Participants) | 41
  Change from BL @ Week 4 | -118.4 (590.20)
  Change from BL @ Week 8: number analyzed (Participants) | 43
  Change from BL @ Week 8 | -17.5 (665.68)
  Change from BL @ Week 12: number analyzed (Participants) | 39
  Change from BL @ Week 12 | -52.8 (790.26)
  Change from BL @ Week 16: number analyzed (Participants) | 42
  Change from BL @ Week 16 | 71.9 (988.30)
  Change from BL @ Week 20: number analyzed (Participants) | 40
  Change from BL @ Week 20 | -64.3 (791.92)
  Change from BL @ EOT (Week 24): number analyzed (Participants) | 39
  Change from BL @ EOT (Week 24) | -140.7 (824.01)

5. Secondary Outcome: Number of Participants With Worst Post-baseline Values in Selected Chemistry Parameters
Description: Safety measured by the worst post-baseline severity grade observed in a patient calculated using the normal/low/high classifications based on local laboratory normal ranges, regardless of the baseline status. Baseline was defined as the last non-missing value on or prior to the first dose. The selected chemistry parameters were: Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Aspartate aminotransferase (AST), total bilirubin, direct bilirubin, serum creatinine and Urine protein creatinine ratio (UPCR) (Protein/Creatinine represented UPCR). Only descriptive analysis performed.
Time Frame: Baseline (Week 1 Day 1) up to Week 24, plus 30 day safety follow-up.
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
Participants
  Alanine Aminotransferase: Normal | 16
  Alanine Aminotransferase: Low | 0
  Alanine Aminotransferase: High | 28
  Alanine Aminotransferase: High & Low | 0
  Alanine Aminotransferase: Missing | 0
  Alkaline Phosphatase: Normal | 25
  Alkaline Phosphatase: Low | 2
  Alkaline Phosphatase: High | 17
  Alkaline Phosphatase: High & Low | 0
  Alkaline Phosphatase: Missing | 0
  Aspartate Aminotransferase: Normal | 14
  Aspartate Aminotransferase: Low | 0
  Aspartate Aminotransferase: High | 30
  Aspartate Aminotransferase: High & Low | 0
  Aspartate Aminotransferase: Missing | 0
  Bilirubin: Normal | 16
  Bilirubin: Low | 0
  Bilirubin: High | 28
  Bilirubin: High & Low | 0
  Bilirubin: Missing | 0
  Creatinine: Normal | 6
  Creatinine: Low | 29
  Creatinine: High | 6
  Creatinine: High & Low | 3
  Creatinine: Missing | 0
  Direct Bilirubin: Normal | 16
  Direct Bilirubin: Low | 0
  Direct Bilirubin: High | 28
  Direct Bilirubin: High & Low | 0
  Direct Bilirubin: Missing | 0
  Protein/Creatinine: Normal | 20
  Protein/Creatinine: Low | 1
  Protein/Creatinine: High | 17
  Protein/Creatinine: High & Low | 6
  Protein/Creatinine: Missing | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Auditory Assessments Changes From Baseline
Description: Safety measured by notable post-baseline changes in Auditory assessments (comprehensive audiometry threshold examination and speech recognition). Baseline was defined as the last non-missing value on or prior to the first dose. Only descriptive analysis performed.
Time Frame: Baseline (Week 1 Day 1) up to Week 24, plus 30 day safety follow-up.
Population: Safety set. For each parameter, only patients with a value at both baseline and post baseline were to be included.
Measure: Number; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
Participants | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Ocular Assessments Changes From Baseline
Description: Safety measured by notable post-baseline changes in Ocular assessments (Distance visual acuity test, Applanation tonometry, lens photography, wide angle fundus photography of the retina and optic nerve). Ocular assessment were required at screening and end of Treatment; during treatment, they were to be performed at the discretion of the investigator based on patient reporting symptoms. Baseline was defined as the last non-missing value on or prior to the first dose. Only descriptive analysis performed.
Time Frame: Baseline (Week 1 Day 1) up to Week 24, plus 30 day safety follow-up.
Population: Safety set. For each parameter, only patients with a value at both baseline and post baseline were to be included.
Measure: Number; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
Participants | 0

8. Secondary Outcome: Absolute Change From Baseline in Systolic and Diastolic Blood Pressures (mmHg)
Description: Absolute change from baseline over time in systolic and diastolic blood pressures measurements were to be provided. Only descriptive analysis performed.
Time Frame: Baseline (BL), Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, EOT (Week 24)
Population: Safety set. For each parameter, only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
millimetre of mercury (mmHg)
  Systolic BP-Baseline (BL) | 100.0 (10.10)
  Systolic BP-Change from BL @ Week 2: number analyzed (Participants) | 37
  Systolic BP-Change from BL @ Week 2 | -0.1 (11.27)
  Systolic BP-Change from BL @ Week 3: number analyzed (Participants) | 38
  Systolic BP-Change from BL @ Week 3 | -2.3 (7.93)
  Systolic BP-Change from BL @ Week 4 | -0.3 (12.56)
  Systolic BP-Change from BL @ Week 8 | 0.3 (8.53)
  Systolic BP-Change from BL @ Week 12: number analyzed (Participants) | 41
  Systolic BP-Change from BL @ Week 12 | -1.4 (12.16)
  Systolic BP-Change from BL @ Week 16: number analyzed (Participants) | 42
  Systolic BP-Change from BL @ Week 16 | -1.9 (11.76)
  Systolic BP-Change from BL @ Week 20: number analyzed (Participants) | 41
  Systolic BP-Change from BL @ Week 20 | -0.6 (11.67)
  Systolic BP-Change from BL @ EOT (Week 24): number analyzed (Participants) | 39
  Systolic BP-Change from BL @ EOT (Week 24) | -2.6 (11.54)
  Diastolic BP-Baseline (BL) | 60.0 (7.85)
  Diastolic BP-Change from BL @ Week 2: number analyzed (Participants) | 37
  Diastolic BP-Change from BL @ Week 2 | 0.7 (6.13)
  Diastolic BP-Change from BL @ Week 3: number analyzed (Participants) | 38
  Diastolic BP-Change from BL @ Week 3 | -2.1 (9.60)
  Diastolic BP-Change from BL @ Week 4 | 1.0 (10.24)
  Diastolic BP-Change from BL @ Week 8 | -0.6 (13.21)
  Diastolic BP-Change from BL @ Week 12: number analyzed (Participants) | 41
  Diastolic BP-Change from BL @ Week 12 | 1.7 (11.42)
  Diastolic BP-Change from BL @ Week 16: number analyzed (Participants) | 42
  Diastolic BP-Change from BL @ Week 16 | -0.5 (10.28)
  Diastolic BP-Change from BL @ Week 20: number analyzed (Participants) | 41
  Diastolic BP-Change from BL @ Week 20 | -0.1 (11.70)
  Diastolic BP-Change from BL @ EOT (Week 24): number analyzed (Participants) | 39
  Diastolic BP-Change from BL @ EOT (Week 24) | -0.4 (7.89)

9. Secondary Outcome: Absolute Change From Baseline in Pulse Rate (Bpm)
Description: Absolute change from baseline over time in supine pulse rate was to be provided. Only descriptive analysis performed.
Time Frame: Baseline (BL), Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, EOT (Week 24)
Population: Safety set. For each parameter, only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
beats per minute (bpm)
  Baseline (BL) | 102.4 (10.73)
  Change from BL @ Week 2: number analyzed (Participants) | 38
  Change from BL @ Week 2 | -1.1 (10.51)
  Change from BL @ Week 3: number analyzed (Participants) | 38
  Change from BL @ Week 3 | -2.7 (16.18)
  Change from BL @ Week 4 | -3.1 (12.85)
  Change from BL @ Week 8 | -1.0 (15.47)
  Change from BL @ Week 12: number analyzed (Participants) | 41
  Change from BL @ Week 12 | -0.3 (12.69)
  Change from BL @ Week 16: number analyzed (Participants) | 42
  Change from BL @ Week 16 | -2.2 (8.99)
  Change from BL @ Week 20: number analyzed (Participants) | 41
  Change from BL @ Week 20 | 0.8 (12.55)
  Change from BL @ EOT (Week 24): number analyzed (Participants) | 39
  Change from BL @ EOT (Week 24) | 1.1 (12.10)

10. Secondary Outcome: Absolute Change From Baseline in Body Temperature (°C)
Description: Absolute change from baseline over time in body temperature measurements was to be provided. Only descriptive analysis performed.
Time Frame: Baseline (BL), Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, EOT (Week 24)
Population: Safety set. For each parameter, only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (Standard Deviation); unit: Celsius degree (°C)
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
Celsius degree (°C)
  Baseline (BL) | 36.43 (0.416)
  Change from BL @ Week 2: number analyzed (Participants) | 38
  Change from BL @ Week 2 | -0.03 (0.285)
  Change from BL @ Week 3: number analyzed (Participants) | 38
  Change from BL @ Week 3 | -0.10 (0.353)
  Change from BL @ Week 4: number analyzed (Participants) | 43
  Change from BL @ Week 4 | 0.00 (0.360)
  Change from BL @ Week 8 | 0.02 (0.336)
  Change from BL @ Week 12: number analyzed (Participants) | 41
  Change from BL @ Week 12 | -0.03 (0.413)
  Change from BL @ Week 16: number analyzed (Participants) | 42
  Change from BL @ Week 16 | 0.10 (0.400)
  Change from BL @ Week 20: number analyzed (Participants) | 41
  Change from BL @ Week 20 | 0.03 (0.372)
  Change from BL @ EOT (Week 24): number analyzed (Participants) | 39
  Change from BL @ EOT (Week 24) | 0.08 (0.453)

11. Secondary Outcome: Absolute Change From Baseline in Body Weight (kg)
Description: Absolute change from baseline over time in body weight measurements was to be provided. Only descriptive analysis performed.
Time Frame: Baseline (BL), Week 4, Week 8, Week 12, Week 16, Week 20, EOT (Week 24)
Population: Safety set. For each parameter, only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Deferasirox
Number analyzed (Participants) | 44
kilogram (kg)
  Baseline (BL) | 15.26 (3.109)
  Change from BL @ Week 4: number analyzed (Participants) | 43
  Change from BL @ Week 4 | 0.08 (0.290)
  Change from BL @ Week 8 | 0.19 (0.460)
  Change from BL @ Week 12: number analyzed (Participants) | 41
  Change from BL @ Week 12 | 0.31 (0.482)
  Change from BL @ Week 16: number analyzed (Participants) | 42
  Change from BL @ Week 16 | 0.25 (0.433)
  Change from BL @ Week 20: number analyzed (Participants) | 41
  Change from BL @ Week 20 | 0.43 (0.532)
  Change from BL @ EOT (Week 24): number analyzed (Participants) | 39
  Change from BL @ EOT (Week 24) | 0.44 (0.600)

12. Secondary Outcome: Modified Satisfaction With Iron Chelation Therapy (Modified SICT) in Participants Pre-treated With Deferasirox: Mean Change From Baseline in Adherence
Description: The mSICT questionnaire was to be completed at screening visit 1, week 4, week 12 and EOT. The responses from screening visit 1 for mSICT questionnaire were to be considered as baseline. The modified SICT consisted of 20 items that represented 3 domains: Adherence, Preference and Concerns. The mSICT adherence domain consisted of 6 items from the child's perspective and 6 items from the caregiver's perspective, each with a possible score of 1 to 5, for an overall possible score range of 6 to 30. A higher score indicates poorer adherence. Only descriptive analysis performed.
Time Frame: Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (95% Confidence Interval); unit: Score
Arm/Group | Deferasirox
Number analyzed (Participants) | 32
Score
  Child's perspective overall score-Week 4: number analyzed (Participants) | 30
  Child's perspective overall score-Week 4 | -2.4 [-3.8 to -1.0]
  Child's perspective overall score-Week 12: number analyzed (Participants) | 27
  Child's perspective overall score-Week 12 | -2.6 [-4.5 to -0.7]
  Child's perspective overall score-EOT: number analyzed (Participants) | 28
  Child's perspective overall score-EOT | -1.9 [-3.5 to -0.2]
  Caregiver's perspective overall score-Week 4: number analyzed (Participants) | 30
  Caregiver's perspective overall score-Week 4 | -1.4 [-2.9 to 0.1]
  Caregiver's perspective overall score-Week 12: number analyzed (Participants) | 27
  Caregiver's perspective overall score-Week 12 | -1.4 [-3.3 to 0.4]
  Caregiver's perspective overall score-EOT: number analyzed (Participants) | 28
  Caregiver's perspective overall score-EOT | -1.0 [-2.6 to 0.6]

13. Secondary Outcome: Modified SICT in Participants Pre-treated With Deferasirox: Number of Participants With Type of Medicine Child Like Scoring
Description: The mSICT questionnaire was to be completed at screening visit 1, week 4, week 12 and EOT. The responses from screening visit 1 for mSICT questionnaire were to be considered as baseline. The modified SICT consisted of 20 items that represented 3 domains: Adherence, Preference and Concerns. The mSICT preference domain consisted of 3 items including the type of medicine the child said he/she liked best (tablet to dissolve in liquid, tablet (taken once a day), tablet (taken 3 times a day), tablet crushed, sprinkle powder on food, injection and I don't know). These items were presented descriptively using frequency counts.
Time Frame: Baseline (BL), Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 32
Participants
  BL: Tablet to dissolve in liquid | 0
  BL: Tablet (taken once a day) | 4
  BL: Tablet (taken 3 times a day) | 0
  BL: Tablet crushed | 11
  BL: Sprinkle powder on food | 14
  BL: Injection | 0
  BL: I don't know | 3
  Wk 4: number analyzed (Participants) | 30
  Wk 4: Tablet to dissolve in liquid | 0
  Wk 4: Tablet (taken once a day) | 1
  Wk 4: Tablet (taken 3 times a day) | 0
  Wk 4: Tablet crushed | 14
  Wk 4: Sprinkle powder on food | 14
  Wk 4: Injection | 0
  Wk 4: I don't know | 1
  Wk 12: number analyzed (Participants) | 27
  Wk 12: Tablet to dissolve in liquid | 1
  Wk 12: Tablet (taken once a day) | 1
  Wk 12: Tablet (taken 3 times a day) | 0
  Wk 12: Tablet crushed | 13
  Wk 12: Sprinkle powder on food | 12
  Wk 12: Injection | 0
  Wk 12: I don't know | 0
  EOT: number analyzed (Participants) | 28
  EOT: Tablet to dissolve in liquid | 0
  EOT: Tablet (taken once a day) | 4
  EOT: Tablet (taken 3 times a day) | 0
  EOT: Tablet crushed | 9
  EOT: Sprinkle powder on food | 15
  EOT: Injection | 0
  EOT: I don't know | 0

14. Secondary Outcome: Modified SICT in Participants Pre-treated With Deferasirox: Number of Participants With Reasons Child Preferred Crushed Medicine Scoring
Description: The mSICT questionnaire was to be completed at screening visit 1, week 4, week 12 and EOT. The responses from screening visit 1 for mSICT questionnaire were to be considered as baseline. The modified SICT consisted of 20 items that represented 3 domains: Adherence, Preference and Concerns. The mSICT preference domain consisted of 3 items including the reason child preferred crushed medicine (taste, aftertaste, convenience, number of pills, no/less side effects, can correctly prepare the medicine, easier to remember to take the medicine, number of times he/she has to take the medicine, no/less pain on the injection site, gain personal time with their family and friends, and other). These items were presented descriptively using frequency counts.
Time Frame: Baseline (BL), Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 32
Participants
  BL: number analyzed (Participants) | 20
  BL: Taste | 6
  BL: Aftertaste | 5
  BL: Convenience | 5
  BL: Number of pills | 0
  BL: No/Less side effects | 0
  BL: Can correctly prepare the medicine | 0
  BL: Easier to remember to take the medicine | 1
  BL: Number of times he/she has to take the medicine | 0
  BL: No/Less pain on the injection site | 0
  BL: Gain personal time with their family and friends | 2
  BL: Other | 1
  Wk 4: number analyzed (Participants) | 14
  Wk 4: Taste | 0
  Wk 4: Aftertaste | 0
  Wk 4: Convenience | 4
  Wk 4: Number of pills | 0
  Wk 4: No/Less side effects | 0
  Wk 4: Can correctly prepare the medicine | 0
  Wk 4: Easier to remember to take the medicine | 0
  Wk 4: Number of times he/she has to take the medicine | 0
  Wk 4: No/Less pain on the injection site | 0
  Wk 4: Gain personal time with their family and friends | 2
  Wk 4: Other | 8
  Wk 12: number analyzed (Participants) | 13
  Wk 12: Taste | 0
  Wk 12: Aftertaste | 0
  Wk 12: Convenience | 2
  Wk 12: Number of pills | 0
  Wk 12: No/Less side effects | 0
  Wk 12: Can correctly prepare the medicine | 0
  Wk 12: Easier to remember to take the medicine | 0
  Wk 12: Number of times he/she has to take the medicine | 0
  Wk 12: No/Less pain on the injection site | 0
  Wk 12: Gain personal time with their family and friends | 3
  Wk 12: Other | 8
  EOT: number analyzed (Participants) | 10
  EOT: Taste | 0
  EOT: Aftertaste | 0
  EOT: Convenience | 0
  EOT: Number of pills | 0
  EOT: No/Less side effects | 0
  EOT: Can correctly prepare the medicine | 0
  EOT: Easier to remember to take the medicine | 0
  EOT: Number of times he/she has to take the medicine | 0
  EOT: No/Less pain on the injection site | 0
  EOT: Gain personal time with their family and friends | 7
  EOT: Other | 3

15. Secondary Outcome: Modified SICT in Participants Pre-treated With Deferasirox: Number of Participants With Rank Based on Child's Preference Scoring
Description: The mSICT questionnaire was to be completed at screening visit 1, week 4, week 12 and EOT. The responses from screening visit 1 for mSICT questionnaire were to be considered as baseline. The modified SICT consisted of 20 items that represented 3 domains: Adherence, Preference and Concerns. The mSICT preference domain consisted of 3 items including the rank of the medicine (tablet to dissolve in liquid, tablet taken once a day, tablet taken 3 times a day, tablet crushed, sprinkle powder on food and injection), with a range of 1 to 6 (1 being most preferred and 6 being least preferred), based on what the child prefers. These items were presented descriptively using frequency count.
Time Frame: Baseline (BL), Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 32
Participants
  BL -Tablet to dissolve in liquid: 1 | 0
  BL -Tablet to dissolve in liquid: 2 | 1
  BL -Tablet to dissolve in liquid: 3 | 12
  BL -Tablet to dissolve in liquid: 4 | 7
  BL -Tablet to dissolve in liquid: 5 | 11
  BL -Tablet to dissolve in liquid: 6 | 1
  Week 4 -Tablet to dissolve in liquid: number analyzed (Participants) | 30
  Week 4 -Tablet to dissolve in liquid: 1 | 0
  Week 4 -Tablet to dissolve in liquid: 2 | 11
  Week 4 -Tablet to dissolve in liquid: 3 | 8
  Week 4 -Tablet to dissolve in liquid: 4 | 3
  Week 4 -Tablet to dissolve in liquid: 5 | 5
  Week 4 -Tablet to dissolve in liquid: 6 | 3
  Week 12-Tablet to dissolve in liquid: number analyzed (Participants) | 26
  Week 12-Tablet to dissolve in liquid: 1 | 1
  Week 12-Tablet to dissolve in liquid: 2 | 7
  Week 12-Tablet to dissolve in liquid: 3 | 7
  Week 12-Tablet to dissolve in liquid: 4 | 4
  Week 12-Tablet to dissolve in liquid: 5 | 7
  Week 12-Tablet to dissolve in liquid: 6 | 0
  EOT-Tablet to dissolve in liquid: number analyzed (Participants) | 28
  EOT-Tablet to dissolve in liquid: 1 | 0
  EOT-Tablet to dissolve in liquid: 2 | 8
  EOT-Tablet to dissolve in liquid: 3 | 8
  EOT-Tablet to dissolve in liquid: 4 | 7
  EOT-Tablet to dissolve in liquid: 5 | 4
  EOT-Tablet to dissolve in liquid: 6 | 1
  BL-Tablet (taken once a day): 1 | 6
  BL-Tablet (taken once a day): 2 | 3
  BL-Tablet (taken once a day): 3 | 15
  BL-Tablet (taken once a day): 4 | 6
  BL-Tablet (taken once a day): 5 | 2
  BL-Tablet (taken once a day): 6 | 0
  Week 4-Tablet (taken once a day): number analyzed (Participants) | 30
  Week 4-Tablet (taken once a day): 1 | 3
  Week 4-Tablet (taken once a day): 2 | 0
  Week 4-Tablet (taken once a day): 3 | 9
  Week 4-Tablet (taken once a day): 4 | 18
  Week 4-Tablet (taken once a day): 5 | 0
  Week 4-Tablet (taken once a day): 6 | 0
  Week 12-Tablet (taken once a day): number analyzed (Participants) | 26
  Week 12-Tablet (taken once a day): 1 | 1
  Week 12-Tablet (taken once a day): 2 | 0
  Week 12-Tablet (taken once a day): 3 | 11
  Week 12-Tablet (taken once a day): 4 | 13
  Week 12-Tablet (taken once a day): 5 | 1
  Week 12-Tablet (taken once a day): 6 | 0
  EOT-Tablet (taken once a day): number analyzed (Participants) | 28
  EOT-Tablet (taken once a day): 1 | 4
  EOT-Tablet (taken once a day): 2 | 0
  EOT-Tablet (taken once a day): 3 | 11
  EOT-Tablet (taken once a day): 4 | 13
  EOT-Tablet (taken once a day): 5 | 0
  EOT-Tablet (taken once a day): 6 | 0
  BL-Tablet (taken 3 times a day): 1 | 0
  BL-Tablet (taken 3 times a day): 2 | 0
  BL-Tablet (taken 3 times a day): 3 | 0
  BL-Tablet (taken 3 times a day): 4 | 14
  BL-Tablet (taken 3 times a day): 5 | 17
  BL-Tablet (taken 3 times a day): 6 | 1
  Week 4-Tablet (taken 3 times a day): number analyzed (Participants) | 30
  Week 4-Tablet (taken 3 times a day): 1 | 0
  Week 4-Tablet (taken 3 times a day): 2 | 1
  Week 4-Tablet (taken 3 times a day): 3 | 1
  Week 4-Tablet (taken 3 times a day): 4 | 6
  Week 4-Tablet (taken 3 times a day): 5 | 21
  Week 4-Tablet (taken 3 times a day): 6 | 1
  Week 12-Tablet (taken 3 times a day): number analyzed (Participants) | 26
  Week 12-Tablet (taken 3 times a day): 1 | 0
  Week 12-Tablet (taken 3 times a day): 2 | 2
  Week 12-Tablet (taken 3 times a day): 3 | 1
  Week 12-Tablet (taken 3 times a day): 4 | 6
  Week 12-Tablet (taken 3 times a day): 5 | 17
  Week 12-Tablet (taken 3 times a day): 6 | 0
  EOT-Tablet (taken 3 times a day): number analyzed (Participants) | 28
  EOT-Tablet (taken 3 times a day): 1 | 0
  EOT-Tablet (taken 3 times a day): 2 | 1
  EOT-Tablet (taken 3 times a day): 3 | 1
  EOT-Tablet (taken 3 times a day): 4 | 3
  EOT-Tablet (taken 3 times a day): 5 | 23
  EOT-Tablet (taken 3 times a day): 6 | 0
  BL-Tablet crushed: 1 | 12
  BL-Tablet crushed: 2 | 14
  BL-Tablet crushed: 3 | 3
  BL-Tablet crushed: 4 | 3
  BL-Tablet crushed: 5 | 0
  BL-Tablet crushed: 6 | 0
  Week 4-Tablet crushed: number analyzed (Participants) | 30
  Week 4-Tablet crushed: 1 | 10
  Week 4-Tablet crushed: 2 | 9
  Week 4-Tablet crushed: 3 | 11
  Week 4-Tablet crushed: 4 | 0
  Week 4-Tablet crushed: 5 | 0
  Week 4-Tablet crushed: 6 | 0
  Week 12-Tablet crushed: number analyzed (Participants) | 26
  Week 12-Tablet crushed: 1 | 8
  Week 12-Tablet crushed: 2 | 9
  Week 12-Tablet crushed: 3 | 6
  Week 12-Tablet crushed: 4 | 2
  Week 12-Tablet crushed: 5 | 0
  Week 12-Tablet crushed: 6 | 1
  EOT-Tablet crushed: number analyzed (Participants) | 28
  EOT-Tablet crushed: 1 | 8
  EOT-Tablet crushed: 2 | 9
  EOT-Tablet crushed: 3 | 8
  EOT-Tablet crushed: 4 | 2
  EOT-Tablet crushed: 5 | 1
  EOT-Tablet crushed: 6 | 0
  BL-Sprinkle powder on food: 1 | 16
  BL-Sprinkle powder on food: 2 | 13
  BL-Sprinkle powder on food: 3 | 1
  BL-Sprinkle powder on food: 4 | 1
  BL-Sprinkle powder on food: 5 | 1
  BL-Sprinkle powder on food: 6 | 0
  Week 4-Sprinkle powder on food: number analyzed (Participants) | 30
  Week 4-Sprinkle powder on food: 1 | 19
  Week 4-Sprinkle powder on food: 2 | 8
  Week 4-Sprinkle powder on food: 3 | 0
  Week 4-Sprinkle powder on food: 4 | 1
  Week 4-Sprinkle powder on food: 5 | 2
  Week 4-Sprinkle powder on food: 6 | 0
  Week 12-Sprinkle powder on food: number analyzed (Participants) | 26
  Week 12-Sprinkle powder on food: 1 | 15
  Week 12-Sprinkle powder on food: 2 | 8
  Week 12-Sprinkle powder on food: 3 | 1
  Week 12-Sprinkle powder on food: 4 | 1
  Week 12-Sprinkle powder on food: 5 | 1
  Week 12-Sprinkle powder on food: 6 | 0
  EOT-Sprinkle powder on food: number analyzed (Participants) | 28
  EOT-Sprinkle powder on food: 1 | 16
  EOT-Sprinkle powder on food: 2 | 10
  EOT-Sprinkle powder on food: 3 | 0
  EOT-Sprinkle powder on food: 4 | 2
  EOT-Sprinkle powder on food: 5 | 0
  EOT-Sprinkle powder on food: 6 | 0
  BL-Injection: 1 | 0
  BL-Injection: 2 | 0
  BL-Injection: 3 | 0
  BL-Injection: 4 | 0
  BL-Injection: 5 | 0
  BL-Injection: 6 | 32
  Week 4-Injection: number analyzed (Participants) | 30
  Week 4-Injection: 1 | 0
  Week 4-Injection: 2 | 0
  Week 4-Injection: 3 | 0
  Week 4-Injection: 4 | 1
  Week 4-Injection: 5 | 1
  Week 4-Injection: 6 | 28
  Week 12-Injection: number analyzed (Participants) | 26
  Week 12-Injection: 1 | 1
  Week 12-Injection: 2 | 0
  Week 12-Injection: 3 | 0
  Week 12-Injection: 4 | 0
  Week 12-Injection: 5 | 0
  Week 12-Injection: 6 | 25
  EOT-Injection: number analyzed (Participants) | 28
  EOT-Injection: 1 | 0
  EOT-Injection: 2 | 0
  EOT-Injection: 3 | 0
  EOT-Injection: 4 | 1
  EOT-Injection: 5 | 0
  EOT-Injection: 6 | 27

16. Secondary Outcome: Modified Satisfaction With Iron Chelation Therapy (Modified SICT) in Participants Pre-treated With Deferasirox: Mean Change From Baseline in Concerns
Description: The mSICT questionnaire was to be completed at screening visit 1, week 4, week 12 and EOT. The responses from screening visit 1 for mSICT questionnaire were to be considered as baseline. The modified SICT consisted of 20 items that represented 3 domains: Adherence, Preference and Concerns. The mSICT concerns domain scale for child's response had a possible range from 2 to 10, based on two questions and the mSICT concerns domain scale for caregiver's responses had the possible range of 1 to 5 based on one question. A higher score indicated fewer concerns. Only descriptive analysis performed.
Time Frame: Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (95% Confidence Interval); unit: Score
Arm/Group | Deferasirox
Number analyzed (Participants) | 32
Score
  Child's perspective overall score-Week 4: number analyzed (Participants) | 30
  Child's perspective overall score-Week 4 | 1.1 [0.6 to 1.7]
  Child's perspective overall score-Week 12: number analyzed (Participants) | 27
  Child's perspective overall score-Week 12 | 1.2 [0.5 to 1.9]
  Child's perspective overall score-EOT: number analyzed (Participants) | 28
  Child's perspective overall score-EOT | 0.8 [0.0 to 1.5]
  Caregiver's perspective overall score-Week 4: number analyzed (Participants) | 30
  Caregiver's perspective overall score-Week 4 | 0.4 [-0.1 to 0.8]
  Caregiver's perspective overall score-Week 12: number analyzed (Participants) | 27
  Caregiver's perspective overall score-Week 12 | 0.4 [-0.2 to 0.9]
  Caregiver's perspective overall score-EOT: number analyzed (Participants) | 28
  Caregiver's perspective overall score-EOT | 0.2 [-0.3 to 0.7]

17. Secondary Outcome: Modified Satisfaction With Iron Chelation Therapy (Modified SICT) in Chelation Naive Participants: Mean Change From Baseline in Adherence
Description: as for outcome 12
Time Frame: Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Deferasirox
Number analyzed (Participants) | 12
Score
  Child's perspective overall score-Week 4: number analyzed (Participants) | 11
  Child's perspective overall score-Week 4 | 10.4 (2.98)
  Child's perspective overall score-Week 12: number analyzed (Participants) | 9
  Child's perspective overall score-Week 12 | 9.8 (2.99)
  Child's perspective overall score-EOT: number analyzed (Participants) | 9
  Child's perspective overall score-EOT | 10.3 (3.43)
  Caregiver's perspective overall score-Week 4: number analyzed (Participants) | 11
  Caregiver's perspective overall score-Week 4 | 9.0 (3.97)
  Caregiver's perspective overall score-Week 12: number analyzed (Participants) | 9
  Caregiver's perspective overall score-Week 12 | 9.9 (5.30)
  Caregiver's perspective overall score-EOT: number analyzed (Participants) | 9
  Caregiver's perspective overall score-EOT | 10.6 (5.03)

18. Secondary Outcome: Modified Satisfaction With Iron Chelation Therapy (Modified SICT) in Chelation Naive Participants: Number of Participants With Type of Medicine Child Like Scoring
Description: as for outcome 13
Time Frame: Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 12
Participants
  Wk 4: number analyzed (Participants) | 11
  Wk 4: Tablet to dissolve in liquid | 0
  Wk 4: Tablet (taken once a day) | 1
  Wk 4: Tablet (taken 3 times a day) | 0
  Wk 4: Tablet crushed | 5
  Wk 4: Sprinkle powder on food | 3
  Wk 4: Injection | 0
  Wk 4: I don't know | 2
  Wk 12: number analyzed (Participants) | 9
  Wk 12: Tablet to dissolve in liquid | 1
  Wk 12: Tablet (taken once a day) | 0
  Wk 12: Tablet (taken 3 times a day) | 0
  Wk 12: Tablet crushed | 5
  Wk 12: Sprinkle powder on food | 3
  Wk 12: Injection | 0
  Wk 12: I don't know | 0
  EOT: number analyzed (Participants) | 9
  EOT: Tablet to dissolve in liquid | 4
  EOT: Tablet (taken once a day) | 0
  EOT: Tablet (taken 3 times a day) | 0
  EOT: Tablet crushed | 3
  EOT: Sprinkle powder on food | 2
  EOT: Injection | 0
  EOT: I don't know | 0

19. Secondary Outcome: Modified Satisfaction With Iron Chelation Therapy (Modified SICT) in Chelation Naive Participants: Number of Participants With Reasons Child Preferred Crushed Medicine Scoring
Description: as for outcome 14
Time Frame: Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 12
Participants
  Wk 4: number analyzed (Participants) | 9
  Wk 4: Taste | 0
  Wk 4: Aftertaste | 1
  Wk 4: Convenience | 2
  Wk 4: Number of pills | 1
  Wk 4: No/Less side effects | 0
  Wk 4: Can correctly prepare the medicine | 1
  Wk 4: Easier to remember to take the medicine | 1
  Wk 4: Number of times he/she has to take the medicine | 1
  Wk 4: No/Less pain on the injection site | 0
  Wk 4: Gain personal time with their family and friends | 1
  Wk 4: Other | 1
  Wk 12: number analyzed (Participants) | 6
  Wk 12: Taste | 0
  Wk 12: Aftertaste | 0
  Wk 12: Convenience | 2
  Wk 12: Number of pills | 0
  Wk 12: No/Less side effects | 0
  Wk 12: Can correctly prepare the medicine | 0
  Wk 12: Easier to remember to take the medicine | 0
  Wk 12: Number of times he/she has to take the medicine | 0
  Wk 12: No/Less pain on the injection site | 1
  Wk 12: Gain personal time with their family and friends | 2
  Wk 12: Other | 1
  EOT: number analyzed (Participants) | 8
  EOT: Taste | 0
  EOT: Aftertaste | 0
  EOT: Convenience | 1
  EOT: Number of pills | 0
  EOT: No/Less side effects | 1
  EOT: Can correctly prepare the medicine | 1
  EOT: Easier to remember to take the medicine | 2
  EOT: Number of times he/she has to take the medicine | 0
  EOT: No/Less pain on the injection site | 1
  EOT: Gain personal time with their family and friends | 2
  EOT: Other | 0

20. Secondary Outcome: Modified Satisfaction With Iron Chelation Therapy (Modified SICT) in Chelation Naive Participants: Number of Participants With Rank Based on Child's Preference Scoring
Description: The mSICT questionnaire was to be completed at screening visit 1, week 4, week 12 and EOT. The responses from screening visit 1 for mSICT questionnaire were to be considered as baseline. The modified SICT consisted of 20 items that represented 3 domains: Adherence, Preference and Concerns. The mSICT preference domain consisted of 3 items including the rank of the medicine (tablet to dissolve in liquid, tablet taken once a day, tablet taken 3 times a day, tablet crushed, sprinkle powder on food and injection), with a range of 1 to 6 (1 being most preferred and 6 being least preferred), based on what the child prefers. These items were presented descriptively using frequency counts.
Time Frame: Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 12
Participants
  Wk 4 -Tablet to dissolve in liquid: number analyzed (Participants) | 10
  Wk 4 -Tablet to dissolve in liquid: 1 | 2
  Wk 4 -Tablet to dissolve in liquid: 2 | 1
  Wk 4 -Tablet to dissolve in liquid: 3 | 2
  Wk 4 -Tablet to dissolve in liquid: 4 | 4
  Wk 4 -Tablet to dissolve in liquid: 5 | 1
  Wk 4 -Tablet to dissolve in liquid: 6 | 0
  Wk 12-Tablet to dissolve in liquid: number analyzed (Participants) | 9
  Wk 12-Tablet to dissolve in liquid: 1 | 2
  Wk 12-Tablet to dissolve in liquid: 2 | 3
  Wk 12-Tablet to dissolve in liquid: 3 | 2
  Wk 12-Tablet to dissolve in liquid: 4 | 0
  Wk 12-Tablet to dissolve in liquid: 5 | 2
  Wk 12-Tablet to dissolve in liquid: 6 | 0
  EOT-Tablet to dissolve in liquid: number analyzed (Participants) | 9
  EOT-Tablet to dissolve in liquid: 1 | 4
  EOT-Tablet to dissolve in liquid: 2 | 2
  EOT-Tablet to dissolve in liquid: 3 | 1
  EOT-Tablet to dissolve in liquid: 4 | 2
  EOT-Tablet to dissolve in liquid: 5 | 0
  EOT-Tablet to dissolve in liquid: 6 | 0
  Wk 4-Tablet (taken once a day): number analyzed (Participants) | 10
  Wk 4-Tablet (taken once a day): 1 | 1
  Wk 4-Tablet (taken once a day): 2 | 3
  Wk 4-Tablet (taken once a day): 3 | 5
  Wk 4-Tablet (taken once a day): 4 | 1
  Wk 4-Tablet (taken once a day): 5 | 0
  Wk 4-Tablet (taken once a day): 6 | 0
  Wk 12-Tablet (taken once a day): number analyzed (Participants) | 9
  Wk 12-Tablet (taken once a day): 1 | 0
  Wk 12-Tablet (taken once a day): 2 | 0
  Wk 12-Tablet (taken once a day): 3 | 2
  Wk 12-Tablet (taken once a day): 4 | 6
  Wk 12-Tablet (taken once a day): 5 | 1
  Wk 12-Tablet (taken once a day): 6 | 0
  EOT-Tablet (taken once a day): number analyzed (Participants) | 9
  EOT-Tablet (taken once a day): 1 | 0
  EOT-Tablet (taken once a day): 2 | 1
  EOT-Tablet (taken once a day): 3 | 3
  EOT-Tablet (taken once a day): 4 | 5
  EOT-Tablet (taken once a day): 5 | 0
  EOT-Tablet (taken once a day): 6 | 0
  Wk 4-Tablet (taken 3 times a day): number analyzed (Participants) | 10
  Wk 4-Tablet (taken 3 times a day): 1 | 1
  Wk 4-Tablet (taken 3 times a day): 2 | 0
  Wk 4-Tablet (taken 3 times a day): 3 | 1
  Wk 4-Tablet (taken 3 times a day): 4 | 3
  Wk 4-Tablet (taken 3 times a day): 5 | 4
  Wk 4-Tablet (taken 3 times a day): 6 | 1
  Wk 12-Tablet (taken 3 times a day): number analyzed (Participants) | 9
  Wk 12-Tablet (taken 3 times a day): 1 | 0
  Wk 12-Tablet (taken 3 times a day): 2 | 1
  Wk 12-Tablet (taken 3 times a day): 3 | 2
  Wk 12-Tablet (taken 3 times a day): 4 | 1
  Wk 12-Tablet (taken 3 times a day): 5 | 5
  Wk 12-Tablet (taken 3 times a day): 6 | 0
  EOT-Tablet (taken 3 times a day): number analyzed (Participants) | 9
  EOT-Tablet (taken 3 times a day): 1 | 0
  EOT-Tablet (taken 3 times a day): 2 | 0
  EOT-Tablet (taken 3 times a day): 3 | 0
  EOT-Tablet (taken 3 times a day): 4 | 0
  EOT-Tablet (taken 3 times a day): 5 | 9
  EOT-Tablet (taken 3 times a day): 6 | 0
  Wk 4-Tablet crushed: number analyzed (Participants) | 10
  Wk 4-Tablet crushed: 1 | 1
  Wk 4-Tablet crushed: 2 | 6
  Wk 4-Tablet crushed: 3 | 1
  Wk 4-Tablet crushed: 4 | 1
  Wk 4-Tablet crushed: 5 | 1
  Wk 4-Tablet crushed: 6 | 0
  Wk 12-Tablet crushed: number analyzed (Participants) | 9
  Wk 12-Tablet crushed: 1 | 1
  Wk 12-Tablet crushed: 2 | 5
  Wk 12-Tablet crushed: 3 | 2
  Wk 12-Tablet crushed: 4 | 0
  Wk 12-Tablet crushed: 5 | 0
  Wk 12-Tablet crushed: 6 | 1
  EOT-Tablet crushed: number analyzed (Participants) | 9
  EOT-Tablet crushed: 1 | 1
  EOT-Tablet crushed: 2 | 4
  EOT-Tablet crushed: 3 | 4
  EOT-Tablet crushed: 4 | 0
  EOT-Tablet crushed: 5 | 0
  EOT-Tablet crushed: 6 | 0
  Wk 4-Sprinkle powder on food: number analyzed (Participants) | 10
  Wk 4-Sprinkle powder on food: 1 | 5
  Wk 4-Sprinkle powder on food: 2 | 0
  Wk 4-Sprinkle powder on food: 3 | 0
  Wk 4-Sprinkle powder on food: 4 | 1
  Wk 4-Sprinkle powder on food: 5 | 3
  Wk 4-Sprinkle powder on food: 6 | 1
  Wk 12-Sprinkle powder on food: number analyzed (Participants) | 9
  Wk 12-Sprinkle powder on food: 1 | 5
  Wk 12-Sprinkle powder on food: 2 | 0
  Wk 12-Sprinkle powder on food: 3 | 1
  Wk 12-Sprinkle powder on food: 4 | 2
  Wk 12-Sprinkle powder on food: 5 | 1
  Wk 12-Sprinkle powder on food: 6 | 0
  EOT-Sprinkle powder on food: number analyzed (Participants) | 9
  EOT-Sprinkle powder on food: 1 | 4
  EOT-Sprinkle powder on food: 2 | 2
  EOT-Sprinkle powder on food: 3 | 1
  EOT-Sprinkle powder on food: 4 | 2
  EOT-Sprinkle powder on food: 5 | 0
  EOT-Sprinkle powder on food: 6 | 0
  Wk 4-Injection: number analyzed (Participants) | 10
  Wk 4-Injection: 1 | 0
  Wk 4-Injection: 2 | 0
  Wk 4-Injection: 3 | 1
  Wk 4-Injection: 4 | 0
  Wk 4-Injection: 5 | 1
  Wk 4-Injection: 6 | 8
  Wk 12-Injection: number analyzed (Participants) | 9
  Wk 12-Injection: 1 | 1
  Wk 12-Injection: 2 | 0
  Wk 12-Injection: 3 | 0
  Wk 12-Injection: 4 | 0
  Wk 12-Injection: 5 | 0
  Wk 12-Injection: 6 | 8
  EOT-Injection: number analyzed (Participants) | 9
  EOT-Injection: 1 | 0
  EOT-Injection: 2 | 0
  EOT-Injection: 3 | 0
  EOT-Injection: 4 | 0
  EOT-Injection: 5 | 0
  EOT-Injection: 6 | 9

21. Secondary Outcome: Modified Satisfaction With Iron Chelation Therapy (Modified SICT) in Chelation Naive Participants: Mean Change From Baseline in Concerns
Description: as for outcome 16
Time Frame: Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Deferasirox
Number analyzed (Participants) | 12
Score
  Child's perspective overall score-Week 4: number analyzed (Participants) | 11
  Child's perspective overall score-Week 4 | 9.7 (0.65)
  Child's perspective overall score-Week 12: number analyzed (Participants) | 9
  Child's perspective overall score-Week 12 | 9.4 (0.88)
  Child's perspective overall score-EOT: number analyzed (Participants) | 9
  Child's perspective overall score-EOT | 8.9 (1.36)
  Caregiver's perspective overall score-Week 4: number analyzed (Participants) | 11
  Caregiver's perspective overall score-Week 4 | 3.7 (1.42)
  Caregiver's perspective overall score-Week 12: number analyzed (Participants) | 9
  Caregiver's perspective overall score-Week 12 | 3.9 (1.76)
  Caregiver's perspective overall score-EOT: number analyzed (Participants) | 9
  Caregiver's perspective overall score-EOT | 3.4 (1.59)

22. Secondary Outcome: Palatability Score in Chelation Naive Participants
Description: The palatability (taste and ability to consume medicine) questionnaire consisted of 4 items, three items measuring taste or ability to consume medicine and one item measuring aftertaste. The aftertaste item was treated separately. Among the taste items, first one measured taste on a five point response scale. The last two items measured what happened after taking the medicine, i.e., swallowed or vomited etc. and how the perceived amount of liquid taken with the medicine was, enough, not enough or too much. The palatability summary score was calculated from these three items using a scoring matrix and the score ranges from 0 to 11. A higher score indicates better palatability. Only descriptive analysis was performed.
Time Frame: Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Deferasirox
Number analyzed (Participants) | 12
Score
  Week 4: number analyzed (Participants) | 10
  Week 4 | 10.4 (0.97)
  Week 12: number analyzed (Participants) | 9
  Week 12 | 10.9 (0.33)
  EOT (Week 24): number analyzed (Participants) | 9
  EOT (Week 24) | 10.8 (0.67)

23. Secondary Outcome: Number of Chelation Naive Participants With Palatability After Taste Item Scoring
Description: The palatability (taste and ability to consume medicine) questionnaire consisted of 4 items, three items measuring taste or ability to consume medicine and one item measuring aftertaste. The aftertaste item was treated as a separate item and scored on a 5-point response scale with the response format Very good = 1 (best), Good = 2, Neither good nor bad = 3, Bad = 4, Very bad = 5 (worst). Only descriptive analysis performed using frequency counts.
Time Frame: Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 12
Participants
  Wk 4: number analyzed (Participants) | 11
  Wk 4: Very Good | 3
  Wk 4: Good | 4
  Wk 4: Neither good nor bad | 3
  Wk 4: Bad | 1
  Wk 4: Very bad | 0
  Wk 12: number analyzed (Participants) | 9
  Wk 12: Very Good | 2
  Wk 12: Good | 5
  Wk 12: Neither good nor bad | 2
  Wk 12: Bad | 0
  Wk 12: Very bad | 0
  EOT: number analyzed (Participants) | 9
  EOT: Very Good | 1
  EOT: Good | 4
  EOT: Neither good nor bad | 3
  EOT: Bad | 1
  EOT: Very bad | 0

24. Secondary Outcome: Palatability Score in Participants Pre-treated With Deferasirox
Description: as for outcome 22
Time Frame: Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Deferasirox
Number analyzed (Participants) | 32
Score
  Week 4: number analyzed (Participants) | 30
  Week 4 | 10.7 (1.29)
  Week 12: number analyzed (Participants) | 27
  Week 12 | 10.3 (2.13)
  EOT (Week 24): number analyzed (Participants) | 28
  EOT (Week 24) | 10.6 (1.57)

25. Secondary Outcome: Number of Participants Pre-treated With Deferasirox With Palatability After Taste Item Scoring
Description: as for outcome 23
Time Frame: Baseline, Week 4, Week 12, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 32
Participants
  BL: Very Good | 5
  BL: Good | 5
  BL: Neither good nor bad | 15
  BL: Bad | 7
  BL: Very bad | 0
  Wk 4: number analyzed (Participants) | 30
  Wk 4: Very Good | 1
  Wk 4: Good | 13
  Wk 4: Neither good nor bad | 16
  Wk 4: Bad | 0
  Wk 4: Very bad | 0
  Wk 12: number analyzed (Participants) | 27
  Wk 12: Very Good | 4
  Wk 12: Good | 9
  Wk 12: Neither good nor bad | 12
  Wk 12: Bad | 2
  Wk 12: Very bad | 0
  EOT: number analyzed (Participants) | 28
  EOT: Very Good | 0
  EOT: Good | 11
  EOT: Neither good nor bad | 14
  EOT: Bad | 3
  EOT: Very bad | 0

26. Secondary Outcome: GI Symptom Score in Chelation Naive Participants
Description: The GI symptom score was calculated from responses to 5 questions, each with a possible score of 1 to 5, for an overall possible score range of 5 to 25, where a lower score represents a less severe GI symptom and a higher score represents a more severe GI symptom. GI symptom scores were summarized using descriptive statistics at week 2, week 3, week 4, week 8, week 12, week 16, week 20 and EOT.
Time Frame: Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Deferasirox
Number analyzed (Participants) | 12
Score
  Week 2 | 6.8 (2.82)
  Week 3: number analyzed (Participants) | 10
  Week 3 | 7.1 (2.85)
  Week 4: number analyzed (Participants) | 11
  Week 4 | 7.0 (3.52)
  Week 8: number analyzed (Participants) | 11
  Week 8 | 6.8 (2.64)
  Week 12: number analyzed (Participants) | 9
  Week 12 | 6.2 (1.79)
  Week 16: number analyzed (Participants) | 9
  Week 16 | 7.0 (2.18)
  Week 20: number analyzed (Participants) | 10
  Week 20 | 5.9 (1.29)
  EOT (Week 24): number analyzed (Participants) | 9
  EOT (Week 24) | 6.8 (1.92)

27. Secondary Outcome: Number of Participants With GI Bowel Movements Item Scoring in Chelation Naive Participants
Description: The GI symptom questionnaire consisted of 6 items, 5 of which were scored using a 1-5 rating scale. The sixth item assessed bowel movement frequency during the past week, using 7 response options 0 = 0 ("None"), 1 = 1, 2 = 2, 3 = 3, 4 = 4, 5 = "5 - 10" and 6 = "11 or more". The GI bowel movements item score was presented descriptively using frequency counts.
Time Frame: Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 12
Participants
  Week 2: 3 | 1
  Week 2: 4 | 1
  Week 2: 5 to 10 | 8
  Week 2: 11 or more | 2
  Week 3: number analyzed (Participants) | 10
  Week 3: 3 | 1
  Week 3: 4 | 0
  Week 3: 5 to 10 | 7
  Week 3: 11 or more | 2
  Week 4: number analyzed (Participants) | 11
  Week 4: 3 | 0
  Week 4: 4 | 1
  Week 4: 5 to 10 | 8
  Week 4: 11 or more | 2
  Week 8: number analyzed (Participants) | 11
  Week 8: 3 | 0
  Week 8: 4 | 3
  Week 8: 5 to 10 | 6
  Week 8: 11 or more | 2
  Week 12: number analyzed (Participants) | 9
  Week 12: 3 | 0
  Week 12: 4 | 2
  Week 12: 5 to 10 | 6
  Week 12: 11 or more | 1
  Week 16: number analyzed (Participants) | 9
  Week 16: 3 | 0
  Week 16: 4 | 2
  Week 16: 5 to 10 | 5
  Week 16: 11 or more | 2
  Week 20: number analyzed (Participants) | 10
  Week 20: 3 | 0
  Week 20: 4 | 1
  Week 20: 5 to 10 | 7
  Week 20: 11 or more | 2
  EOT (Week 24): number analyzed (Participants) | 9
  EOT (Week 24): 3 | 2
  EOT (Week 24): 4 | 0
  EOT (Week 24): 5 to 10 | 6
  EOT (Week 24): 11 or more | 1

28. Secondary Outcome: GI Symptom Score in Participants Pre-treated With Deferasirox
Description: as for outcome 26
Time Frame: Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Deferasirox
Number analyzed (Participants) | 32
Score
  Week 2 | 6.3 (1.91)
  Week 3: number analyzed (Participants) | 28
  Week 3 | 6.0 (1.63)
  Week 4: number analyzed (Participants) | 30
  Week 4 | 6.4 (1.81)
  Week 8 | 6.4 (2.34)
  Week 12: number analyzed (Participants) | 27
  Week 12 | 6.5 (1.83)
  Week 16: number analyzed (Participants) | 31
  Week 16 | 6.7 (2.10)
  Week 20: number analyzed (Participants) | 31
  Week 20 | 7.3 (2.37)
  EOT (Week 24): number analyzed (Participants) | 28
  EOT (Week 24) | 7.6 (2.95)

29. Secondary Outcome: Number of Participants With GI Bowel Movements Item Scoring in Participants Pre-treated With Deferasirox
Description: as for outcome 27
Time Frame: Baseline, Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, EOT (Week 24)
Population: Full Analysis Set (FAS). Only patients with a value at both baseline and post baseline were to be included.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 32
Participants
  Baseline (BL): 3 | 0
  Baseline (BL): 4 | 1
  Baseline (BL): 5 to 10 | 30
  Baseline (BL): 11 or more | 1
  Week 2: 3 | 0
  Week 2: 4 | 1
  Week 2: 5 to 10 | 29
  Week 2: 11 or more | 2
  Week 3: number analyzed (Participants) | 28
  Week 3: 3 | 0
  Week 3: 4 | 1
  Week 3: 5 to 10 | 26
  Week 3: 11 or more | 1
  Week 4: number analyzed (Participants) | 30
  Week 4: 3 | 0
  Week 4: 4 | 1
  Week 4: 5 to 10 | 28
  Week 4: 11 or more | 1
  Week 8: 3 | 1
  Week 8: 4 | 1
  Week 8: 5 to 10 | 29
  Week 8: 11 or more | 1
  Week 12: number analyzed (Participants) | 27
  Week 12: 3 | 1
  Week 12: 4 | 0
  Week 12: 5 to 10 | 26
  Week 12: 11 or more | 0
  Week 16: number analyzed (Participants) | 31
  Week 16: 3 | 0
  Week 16: 4 | 1
  Week 16: 5 to 10 | 29
  Week 16: 11 or more | 1
  Week 20: number analyzed (Participants) | 31
  Week 20: 3 | 0
  Week 20: 4 | 1
  Week 20: 5 to 10 | 28
  Week 20: 11 or more | 2
  EOT (Week 24): number analyzed (Participants) | 28
  EOT (Week 24): 3 | 0
  EOT (Week 24): 4 | 1
  EOT (Week 24): 5 to 10 | 25
  EOT (Week 24): 11 or more | 2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from first dose of study treatment until end of study treatment plus 30 days post-treatment, assessed for approximately 28 weeks.
Description: Any sign or symptom that occurs during the study treatment and 30 days post treatment follow up. Maximum exposure to study treatment = 26 weeks
Arm/Group | Deferasirox
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 2/44
Other Adverse Events (participants affected / at risk) | 29/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=44)
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=44)
Diarrhoea (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 5
Gastroenteritis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 10
Alanine aminotransferase increased (Investigations) | 7
Bilirubin conjugated increased (Investigations) | 6
Blood creatinine increased (Investigations) | 9
Urine protein/creatinine ratio increased (Investigations) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT03372083/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT03372083/SAP_001.pdf